CLINICAL TRIAL: NCT05990868
Title: Administration of Rectal Acetaminophen During Oocyte Retrievals Reduces Post-Operative Opioid Utilization in Fertility Patients.
Brief Title: Rectal Acetaminophen During Oocyte Retrievals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Anthony Imudia, Associate Professor, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY005325
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Oocyte Retrieival and Post Operative Pain Control
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: The primary outcome in this study is the proportion of the prescribed medications used three days after discharge from the surgery. Assuming that only one third or less of the Narcotics prescribed (2 out of 6 tablets) in Group 1 will be utilized as compared to two thirds or more (4 out of 6 tables) in group 2, 35 patients in each group will be required to achieve 80% power and two-sided level of significance of 0.058. Given we expect possible 10% drop out rate after randomization, we plan to recruit 39 patients in each group (78 total sample). We plan to perform our analysis using SPSS.
Who Masked: Participant, Care Provider
Masking Description: Both patient and provider will be blinded to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rectal tylenol group: Group 1 (Active Comparator): Randomization to the study group (Group 1): will receive standard anesthesia and 650 mg rectal Tylenol at the time of egg retrieval.
  Interventions: Drug: Tylenol
- Placebo group: Group 2 (Placebo Comparator): Randomization to the standard of care group (Group 2): will receive standard anesthesia and rectal placebo at the time of oocyte retrieval. Placebo is a substance that has no therapeutic effect and used as a control in testing new drugs.
  Interventions: Drug: Tylenol

INTERVENTIONS:
Drug: Tylenol — Rectal tylenol will be placed at the time of oocyte retrieval

SUMMARY:
As the opioid epidemic shows no sign of abating, this national crisis deserves careful attention from all medical subspecialties. This includes reproductive endocrinology and infertility (REI), where opioids are primarily utilized for intraoperative and postoperative pain management for outpatient procedures such as oocyte retrievals, operative hysteroscopy, and laparoscopic myomectomy. The primary aim of this study is to evaluate whether or not the administration of rectal acetaminophen as an alternative analgesic at the completion of oocyte retrieval would reduce postoperative utilization of opioids (Tylenol with oxycodone) in fertility patients. This trial has the potential to provide practice-changing clinical information to the field of REI. The information gained can even translate to other ambulatory procedures and guide clinical practice.

Primary objective of the study will be to identify the proportion of prescribed Acetaminophen and Narcotics utilized 3 days following oocyte retrieval.

DETAILED DESCRIPTION:
There are various methods of anesthesia used for transvaginal ultrasound guided oocyte retrievals. The majority of cases are performed under conscious sedation with a combination of sedative-hypnotic agents and analgesics while a small proportion of these retrievals are performed under general, regional, or local anesthesia. Conscious sedation is defined as, "a minimally depressed level of consciousness that retains the patient's ability to maintain a patent airway independently and continuously and to respond appropriately to physical stimulation and verbal commands."1 The most common agents chosen for conscious sedation are midazolam and/or Propofol with fentanyl for analgesia in some cases. One retrospective study looking at over a thousand patients undergoing oocyte retrieval at an in vitro fertilization (IVF) center found that no complications developed relating to anesthesia. Several cross-sectional studies looking at patients undergoing ultrasound-guided transvaginal follicle aspiration found that there was high patient satisfaction with a conscious sedation protocol of midazolam and opioid analgesia. Although this technique of conscious sedation has been the standard of care for several decades demonstrating good patient satisfaction and complications are rare, patients are still given oral opioids for postoperative pain. Given current opioid addiction crisis, it is prudent to challenge current practice by evaluating possible interventions that could help reduce both intraoperative and postoperative administration of opioids to fertility patients.

The pain experienced in oocyte retrieval is caused by the needle puncturing through the vaginal wall and by the mechanical stimulation of the ovary. This pain is often described as similar to intense menstrual cramping4. The retrospective study referenced above evaluated patients' self-reported degrees of pain and found that over 80% of patients undergoing oocyte retrieval reported having only mild pain or no pain at all5. Another study found that 6.9% of patients undergoing oocyte retrieval reported the procedure to be very or extremely painful with significant predictors of pain being negative gynecological experiences, having experienced side effects during their hormonal treatment, higher levels of intraoperative anxiety, lower levels of perceived control, and longer duration of the retrieval procedure.

Given that most patients seem to tolerate the procedure well, this is a potential clinical area in which opioid use could be minimized, or even eliminated, and non-opioid analgesia could be employed instead.

The current opioid addiction epidemic is one that has been called the "most consequential preventable public health problem in the United States." Although the in-vitro fertilization demographic is not typically associated with substance abuse, it is thought that about six percent of opioid naïve patients are at an increased risk for abusing the medication after surgery and developing new persistent opioid use after being prescribed opioids after an elective surgical procedure. In a study by Bortelleto et al it was reported that approximately 12 % of women fill up opioid prescription after oocyte retrieval8. In a recent study by Petrozza et al evaluated use of IV Acetaminophen in oocyte retrieval and reported that preoperative IV acetaminophen did not reduce postoperative pain scores or shorten the time to discharge when compared with PO acetaminophen or placebo and, thus, cannot currently be recommended routinely in this patient population. Thus, the purpose of this study is to evaluate whether intra-procedure administration of rectal Acetaminophen would be sufficient to manage postoperative pain after oocyte retrievals and could help decrease utilization of prescribed opioid at home following oocyte retrieval.

The primary outcome of this study is to determine the proportion of prescribed Acetaminophen and Opioids (oxycodone) used for the management of pain 3 days after egg retrieval.

ELIGIBILITY:
Inclusion Criteria: Any female patient undergoing oocyte retrieval by transvaginal ultrasound-guided ovarian puncture.

-

Exclusion Criteria:

1. Patients with chronic pain conditions such as fibromyalgia and sickle cell anemia.
2. Patient with BMI greater than 40
3. Patients undergoing transabdominal ultrasound guided oocyte retrieval
4. Patients that required general endotracheal intubation anesthesia in prior oocyte retrieval.
5. Patients with documented allergic reaction to acetaminophen or oxycodone
6. Patient with contra-indication to the use of acetaminophen (liver disease)
7. Patients with a history of past or current alcohol, drug or opioid abuse.
8. Patients with ulcerative colitis, Crohn's disease, or severe rectal hemorrhoids.
9. Patients who develop complication such as PID post procedure.

   -

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only females can undergo oocyte retrieval as they are the gender with ovaries. Our study involves oocyte retrieval procedure.
Enrollment: 78 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Evaluate reduction in opioid use post oocyte retrieval | 1 year
  to determine the proportion of prescribed Acetaminophen and Opioids (oxycodone) used for the management of pain 3 days after egg retrieval.

IPD SHARING:
Plan to Share IPD: Undecided